CLINICAL TRIAL: NCT03661905
Title: Enhancing the Acceptability of Psychological Treatments for Obsessive-compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Collaborators: Université de Montréal (Other); McGill University (Other); University of British Columbia (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Adam S. Radomsky, Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30006258
Record Dates: First submitted 2018-08-20; First posted 2018-09-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Treatment acceptability; Cognitive therapy; Anxiety disorders
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A two-arm parallel assignment where one group will receive Cognitive therapy, and the other group will receive ERP.
Who Masked: Outcomes Assessor
Masking Description: Intervention assessors will not know which participants have been assigned to the different interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Therapy (Experimental): A modularized, cognitive-behavioural therapy intervention that incorporates evidence gathering and behavioural experiments. Our CT protocols rely heavily on behavioural experiments which are typically targeted and brief exercises designed to permit clients/patients to gather disconfirmatory evidence about their beliefs.
  Interventions: Other: Cognitive therapy
- Behavioural Therapy (Active Comparator): Method of behavioral therapy and form of exposure and response prevention therapy in which individuals confront their fears and discontinue their escape response. Exposures in this protocol are prolonged and repeated, requiring clients/patients to engage in a series of exposures to feared stimuli (e.g., contaminants, doubts, intrusive thoughts), and to refrain from engaging in compulsive behaviour until their anxiety subsides.
  Interventions: Behavioral: Exposure and Response Prevention

INTERVENTIONS:
Other: Cognitive therapy — Empirically-supported psychological intervention for various mental health concerns including obsessive-compulsive disorder (OCD). Twelve treatment sessions include components to foster cognitive (i.e. thinking) and behavioural changes.
  Arms: Cognitive Therapy
Behavioral: Exposure and Response Prevention — Exposure therapy in which individuals confront their fears and discontinue their escape response. Twelve treatment sessions implementing exposure which is prolonged and repeated, requiring clients/patients to engage in a series of exposures to feared stimuli (e.g., contaminants, doubts, intrusive thoughts), and to refrain from engaging in compulsive behaviour until their anxiety subsides.
  Arms: Behavioural Therapy

SUMMARY:
Effective treatments for obsessive-compulsive disorder (OCD) usually emphasize a behavioural approach called Exposure and Response Prevention (ERP). In this treatment, patients are encouraged to face their fears repeatedly and for extended periods of time, with the help and support of a caring therapist. Although this is an approach that has been shown to work, many patients find the treatment to be difficult; some even refuse the treatment, or drop out before improvements are seen. The investigators have been working to develop an alternate approach which is just as effective as ERP, but which the investigators think will be much more acceptable to those who seek help for their OCD. This study will compare the traditional behavioural approach, with the newer cognitively-based approach. The investigators expect that the two treatments will both reduce the symptoms and distress of people with OCD, but that this newer cognitive therapy will have fewer people who refuse or drop out of the treatment, and will be rated as more acceptable. This research will have important implications not only for those struggling with OCD, but also for other anxiety-related problems where behavioural approaches are typically recommended, including posttraumatic stress disorder, social anxiety disorder, and other problems.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a serious and often severe mental disorder and one of the leading causes of disability worldwide. Effective psychological interventions for OCD exist, but the prevailing option (Exposure and Response Prevention; ERP) has changed very little since it was established in the 1960's; moreover, it is associated with unacceptably high numbers of individuals who drop out from, or refuse the treatment altogether. This is largely because ERP is a difficult treatment, wherein individuals face their fears with increasing difficulty over time. Just as with the development from early chemotherapy and HIV agents, which were effective, but associated with serious and often severe side effects, it is now time to enhance the acceptability of psychological treatments for OCD.

A novel cognitive therapy (CT) approach is likely to be just as effective as ERP, but markedly more acceptable to those who need it. Although CT for OCD is as effective as ERP, previously tested CTs have failed to incorporate recent experimental research, novel cognitive targets or enhancements to acceptability. Indeed, the investigators recent work on treatment acceptability promises to increase the number of individuals who can fully and successfully engage with the treatment.

The purpose of this research is to enhance the acceptability of cognitive-behavioural treatments for OCD; the investigators aim to accomplish this via a randomized controlled trial comparing traditional ERP against the investigators' novel CT approach. Although the investigators expect both treatments to be effective, the primary hypothesis is that CT will be significantly more acceptable to participants than ERP; this will be assessed by the relative numbers of treatment refusers and dropouts, as well as by participant ratings of treatment acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD
* Ability to read, write, and communicate in English

Exclusion Criteria:

* Psychosis
* Diagnosis of bipolar disorder (I or II)
* Current suicidal ideation/intent
* Current substance abuse
* If participants are on medication they must be on a stable dose (i.e. have maintained a consistent dose for at least three months) and agree not to change their medication regimen for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-26 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidents of participants that drop-out of treatment | Week 2, through treatment completion.
  The investigators will keep a record of the number of participants that drop-out of treatment.
Incidents of participants that refuse treatment | Baseline, up to week two.
  The investigators will keep a record of the number of participants that refuse the treatment.
Treatment and Acceptability Adherence Scale (TAAS; Milosevic, Levy, Alcolado & Radomsky, 2015) | Through study completion (week 3; week 6; one week post therapy; 6 month follow-up; 12 month follow-up).
  The TAAS is a validated 10-item self-report questionnaire designed to assess treatment acceptability and anticipated adherence in response to a given treatment for anxiety and related problems. It is intended to be administered to potential treatment recipients after they have received information about the treatment. Items are rated on a 7-point Likert-type scale (1 Disagree strongly; 7 Agree strongly) to assess the degree to which participants agree with a variety of statements about a given treatment. Total scores are obtained by summing across all items after negatively worded items (3, 4, 5, 7, 8 and 10) have been reverse-scored. Scores may range from 10 to 70, with higher scores indicating greater acceptability of treatment and greater anticipated ability to adhere to it.

SECONDARY OUTCOMES:
The Vancouver Obsessional Compulsive Inventory (VOCI; Thordarson, Radomsky, Rachman, et al., 2004) | Through study completion (Baseline; week 6; one week post therapy; 6 month follow-up; 12 month follow-up).
  The VOCI is a 55-item self-report scale designed to assess obsessive-compulsive symptom severity. It includes six subscales assessing various symptoms associated with OCD: checking; contamination; obsessions; just right; indecisiveness; and hoarding. Items are rated on a 5-point Likert-type scale (0 Not at all; 4 Very much), with higher scores indicating higher symptom severity.
Anxiety Disorders Interview Schedule for DSM-5 (ADIS-5; Brown & Barlow, 2014) | Through study completion (Baseline; one week post therapy; 6 month follow-up; 12 month follow-up).
  A semi structured diagnostic interview for anxiety disorders and selected other problems (e.g., depression, substance-related disorders). It assesses a variety of current and lifetime symptoms associated with anxiety and other (e.g., mood, somatoform, substance abuse, psychotic) disorders, according to DSM-V criteria.
The Yale-Brown Obsessive Compulsive Scale (YBOCS; Goodman, Price, Rasmussen, et al., 1989) | Through study completion (Baseline; week 6; one week post therapy; 6 month follow-up; 12 month follow-up).
  This 10-item clinician-administered validated measure consists of two subscales, which assess the severity of participants' obsessions and compulsions and monitors symptom improvement during treatment. Subscale scores are summed with a range from 0 (no symptoms) to 40 (severe OCD), with a score less than 8 considered as subclinical symptomatology, over 16 as clinically significant symptoms, and over 24 as moderate to severe OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Radomsky, PhD, Principal Investigator — Concordia University, Montreal
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03661905/Prot_SAP_000.pdf